CLINICAL TRIAL: NCT03359538
Title: Rapamycin (Sirolimus) Treatment for Amyotrophic Lateral Sclerosis
Brief Title: Rapamycin Treatment for ALS
Acronym: RAP-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other); University of Turin, Italy (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Azienda Ospedaliera Niguarda Cà Granda (Other); Fondazione Salvatore Maugeri (Other); University of Padova (Other)
Responsible Party: Principal Investigator, JESSICA MANDRIOLI, MD, PI, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAP-ALS
Record Dates: First submitted 2017-11-08; First posted 2017-12-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Rapamycin
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: treatment double blinded to patients and physicians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator): Patients assigned to this arm will take Riluzole as usual + placebo tablets
  Interventions: Drug: Placebo Oral Tablet
- Rapamycin 1 mg/m2 (Active Comparator): Patients assigned to this arm will take Riluzole as usual + tablets corresponding to a Rapamycin dose of 1 mg/m2/day
  Interventions: Drug: Rapamycin; Drug: Placebo Oral Tablet
- Rapamycin 2 mg/m2 (Active Comparator): Patients assigned to this arm will take Riluzole as usual + tablets corresponding to a Rapamycin dose of 2 mg/m2/day
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — tablets containing Rapamycin/placebo will be administered based on body surface area and adjusted taking into consideration plasma rapamycin dosage
  Other Names: Rapamune
  Arms: Rapamycin 1 mg/m2; Rapamycin 2 mg/m2
Drug: Placebo Oral Tablet — tablets containing Rapamycin/placebo will be administered based on body surface area and adjusted taking into consideration plasma rapamycin dosage
  Arms: Rapamycin 1 mg/m2; placebo

SUMMARY:
In the last years research has pointed out potential mechanisms of pathogenesis in ALS including lack of degradation of abnormally accumulated proteins inside motor neurons, and an unbalanced function of the immune system leading to the prevalence of a neurotoxic function over neuroprotection. These two mechanisms contribute to ALS progression hence representing important therapeutic targets to modify disease expression.

With a phase II clinical trial the investigators aim to study the biological response in ALS treated with Rapamycin, to obtain predictive information for a larger study.

Eight Italian Centres will enroll 63 patients; treatment will be double blinded to patients and physicians, and will last 18 weeks.Follow up will be carried out for 36 months (total duration: 54 weeks).

DETAILED DESCRIPTION:
This is a phase II randomized, double-blind, placebo-controlled, multicenter clinical trial for people with ALS.

The aim is to study the biological and clinical effect of Rapamycin (in two different doses) in addition to Riluzole on ALS patients through comparison with patients treated with Riluzole and placebo.

Rapamycin has been shown to enhance proteins degradation, and this has been associated with beneficial effects in models of neurodegeneration. Its immunomodulatory effects are also well established, notably the ability to suppress inflammatory neurotoxic responses mediated by T cells. As ALS is characterized by heterogeneous pathology and protein accumulation, some patients may respond to therapies that accelerate the clearance of abnormally accumulated proteic aggregates, while suppressing neurotoxic immune elements.

Subjects will be enrolled in 3 groups of 21 subjects; treatment will be double blinded to patients and physicians, and will last 18 weeks. Active treatment will include oral Rapamycin at different doses: Rapamycin 1mg/m2/day or Rapamycin 2mg/m2/day. Rapamycin will be administered at fast, in the morning, once a day. Rapamycin levels will be measured (HPLC) to avoid toxicity (>15 ng/ml), but treating neurologists will have no access to blood laboratory data. Dosages will be adjusted accordingly and sham adjustments will be done in the placebo Group too. Post-treatment follow up will be 36 weeks. Globally the study will lasts 24 months. To monitor adverse events, examination and routine laboratory work (cell count, lipids and protein profile, kidney and liver function, C reactive protein) will be performed before taking Rapamycin/placebo. Non-routine laboratory studies include quantification and characterization of Tregs, lymphocytes phenotype, mTOR (mammilian target of rapamycin) downstream pathway activation in peripheral blood mononuclear cells (PBMC), inflammasome components in PBMC and proinflammatory cytokine production in monocytes, peripheral biomarkers. Cerebrospinal fluid (CSF) will be taken at baseline and at week 18 to measure neurofilaments and to dose Rapamycin to understand whether sufficient levels of Rapamycin can be found in the central nervous system (CNS).

ELIGIBILITY:
Inclusion criteria:

* Patient diagnosed with a laboratory supported , clinically "probable" or "definite" amyotrophic lateral sclerosis according to the Revised El Escorial criteria (Brooks, 2000)
* Familial or sporadic ALS
* Female or male patients aged between 18 and 75 years old
* Disease duration from symptoms onset no longer than 18 months at the screening visit
* Patient treated with a stable dose of Riluzole (100 mg/day) for at least 30 days prior to screening
* Patients with a weight > 50 kg and a BMI ≥18
* Patient with a FVC ≥ 70 % predicted normal value for gender, height, and age at the screening visit
* Patient able and willing to comply with study procedures as per protocol
* Patient able to understand, and capable of providing informed consent at screening visit prior to any protocol-specific procedures
* Use of effective contraception both for males and females

Exclusion Criteria:

* Prior use of Sirolimus
* Prior allergy/sensitivity to Sirolimus or macrolides
* Any medical disorder that would make immunosuppression contraindicated, including but not limited to, acute infections requiring antibiotics, patients with known diagnosis of HIV, tuberculosis, hepatitis B or C infection or history of malignancy
* Severe comorbidities (heart, renal, liver failure), autoimmune diseases or any type of interstitial lung disease
* White blood cells<4,000/mm³, platelets count<100,000/mm³, hematocrit<30%
* Patient who underwent non invasive ventilation, tracheotomy and /or gastrostomy
* Women who are pregnant or breastfeeding
* Participation in pharmacological studies within the last 30 days before screening
* Patients with known superoxide dismutase 1 (SOD1) mutation or with familial ALS and a family member carrying SOD1 mutation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
T-reg number | comparison between baseline and treatment end (week 18)
  Proportion of patients exhibiting a positive response (considered as increase in Treg of at least 30%), comparing baseline and treatment end between Rapamycin and placebo arm

SECONDARY OUTCOMES:
Number of serious adverse events (SAEs) and AEs in placebo and treatment arms | At week 18 and 54
  Rapamycin safety and tolerability in a cohort of ALS patients
Rapamycin capacity to pass through blood brain barrier | At week 18
  HPLC-MS (mass spectrometry) dosage of Rapamycin in CSF in placebo and treatment arm will be performed at treatment end
Rapamycin efficacy in inhibiting Mtor pathway | At week 8-18-30-54
  Assessment of the phosphorylation of the S6 ribosomal protein (S6RP) comparing Rapamycin arms and placebo arm
Changes in activation and homing capabilities of different T, B, natural killer (NK) cell subpopulations | At baseline and at week 8-18-30-54
  Change from baseline to each time point (week 8, 18, 30, and 54) of the activation and homing capabilities of different T, B, NK cell subpopulations comparing Rapamycin arms and placebo arm.
Changes in CSF neurofilaments | Baseline and week 18
  Changes from baseline to week 18 of the levels of neurofilaments in CSF in treatment and placebo arms
Changes in blood biomarkers | Baseline, week 8-18-30-54
  Changes from baseline to week 8-18-30.54 of the levels of neurofilaments and vitamin D in treatment and placebo arms
Rapamycin-induced changes in inflammatory status | Baseline and week 8-18-30-54
  Changes from baseline to each time point (week 8, 18, 30, and 54) in inflammatory status (cytokines and cells) (molecular analysis of the inflammasome system) comparing Rapamycin arms and placebo arm
Changes in Amyotrophic Lateral Sclerosis functional rating scale (ALSFRS)-Revised | Up to week 54
  ALSFRS-R score changes from baseline to week 4, 8, 12, 18, 30, 42 and week 54 in treatment and placebo arms.
Tracheostomy-free survival rate | Up to week 54
  Overall survival from randomization to date of death or tracheostomy
Changes in Forced vital capacity (FVC) | Up to week 54
  Changes in FVC score from baseline to week 4, 8, 12, 18, 30, 42, 54 in treatment and placebo arms.
Change in quality of life | From baseline to week 8, 18, 30 and week 54
  Changes in Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) from baseline to week 8, 18, 30 and week 54, in placebo and treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Mandrioli, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena
Locations (7):
- Italy (7):
  - Centro Sla, Irccs A.O.U. S.Martino Ist, Genova, Genova
  - Centro Clinico Nemo, Fondazione Serena Onlus, Milano, Milan
  - Centro Sla, Irccs Istituto Carlo Besta, Milano, Milan
  - Centro Sla, Ospedale Civile S. Agostino Estense, A.O.U. Modena, Modena
  - Centro Sla, A.O.U. Maggiore Della Carita', Novara, Novara
  - Centro Sla, Universita' Di Padova, Padua
  - Centro Sla, Universita' Di Torino, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barmada SJ, Serio A, Arjun A, Bilican B, Daub A, Ando DM, Tsvetkov A, Pleiss M, Li X, Peisach D, Shaw C, Chandran S, Finkbeiner S. Autophagy induction enhances TDP43 turnover and survival in neuronal ALS models. Nat Chem Biol. 2014 Aug;10(8):677-85. doi: 10.1038/nchembio.1563. Epub 2014 Jun 29. PMID 24974230
- [Background] Beers DR, Henkel JS, Zhao W, Wang J, Huang A, Wen S, Liao B, Appel SH. Endogenous regulatory T lymphocytes ameliorate amyotrophic lateral sclerosis in mice and correlate with disease progression in patients with amyotrophic lateral sclerosis. Brain. 2011 May;134(Pt 5):1293-314. doi: 10.1093/brain/awr074. PMID 21596768
- [Background] Buchan JR, Kolaitis RM, Taylor JP, Parker R. Eukaryotic stress granules are cleared by autophagy and Cdc48/VCP function. Cell. 2013 Jun 20;153(7):1461-74. doi: 10.1016/j.cell.2013.05.037. PMID 23791177
- [Background] Caccamo A, Majumder S, Deng JJ, Bai Y, Thornton FB, Oddo S. Rapamycin rescues TDP-43 mislocalization and the associated low molecular mass neurofilament instability. J Biol Chem. 2009 Oct 2;284(40):27416-24. doi: 10.1074/jbc.M109.031278. Epub 2009 Aug 3. PMID 19651785
- [Background] Chio A, Hammond ER, Mora G, Bonito V, Filippini G. Development and evaluation of a clinical staging system for amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2015 Jan;86(1):38-44. doi: 10.1136/jnnp-2013-306589. Epub 2013 Dec 13. PMID 24336810
- [Background] Cirulli ET, Lasseigne BN, Petrovski S, Sapp PC, Dion PA, Leblond CS, Couthouis J, Lu YF, Wang Q, Krueger BJ, Ren Z, Keebler J, Han Y, Levy SE, Boone BE, Wimbish JR, Waite LL, Jones AL, Carulli JP, Day-Williams AG, Staropoli JF, Xin WW, Chesi A, Raphael AR, McKenna-Yasek D, Cady J, Vianney de Jong JM, Kenna KP, Smith BN, Topp S, Miller J, Gkazi A; FALS Sequencing Consortium; Al-Chalabi A, van den Berg LH, Veldink J, Silani V, Ticozzi N, Shaw CE, Baloh RH, Appel S, Simpson E, Lagier-Tourenne C, Pulst SM, Gibson S, Trojanowski JQ, Elman L, McCluskey L, Grossman M, Shneider NA, Chung WK, Ravits JM, Glass JD, Sims KB, Van Deerlin VM, Maniatis T, Hayes SD, Ordureau A, Swarup S, Landers J, Baas F, Allen AS, Bedlack RS, Harper JW, Gitler AD, Rouleau GA, Brown R, Harms MB, Cooper GM, Harris T, Myers RM, Goldstein DB. Exome sequencing in amyotrophic lateral sclerosis identifies risk genes and pathways. Science. 2015 Mar 27;347(6229):1436-41. doi: 10.1126/science.aaa3650. Epub 2015 Feb 19. PMID 25700176
- [Background] Cloughesy TF, Yoshimoto K, Nghiemphu P, Brown K, Dang J, Zhu S, Hsueh T, Chen Y, Wang W, Youngkin D, Liau L, Martin N, Becker D, Bergsneider M, Lai A, Green R, Oglesby T, Koleto M, Trent J, Horvath S, Mischel PS, Mellinghoff IK, Sawyers CL. Antitumor activity of rapamycin in a Phase I trial for patients with recurrent PTEN-deficient glioblastoma. PLoS Med. 2008 Jan 22;5(1):e8. doi: 10.1371/journal.pmed.0050008. PMID 18215105
- [Background] Deivasigamani S, Verma HK, Ueda R, Ratnaparkhi A, Ratnaparkhi GS. A genetic screen identifies Tor as an interactor of VAPB in a Drosophila model of amyotrophic lateral sclerosis. Biol Open. 2014 Oct 31;3(11):1127-38. doi: 10.1242/bio.201410066. PMID 25361581
- [Background] Harrison DE, Strong R, Sharp ZD, Nelson JF, Astle CM, Flurkey K, Nadon NL, Wilkinson JE, Frenkel K, Carter CS, Pahor M, Javors MA, Fernandez E, Miller RA. Rapamycin fed late in life extends lifespan in genetically heterogeneous mice. Nature. 2009 Jul 16;460(7253):392-5. doi: 10.1038/nature08221. Epub 2009 Jul 8. PMID 19587680
- [Background] Kimura F, Fujimura C, Ishida S, Nakajima H, Furutama D, Uehara H, Shinoda K, Sugino M, Hanafusa T. Progression rate of ALSFRS-R at time of diagnosis predicts survival time in ALS. Neurology. 2006 Jan 24;66(2):265-7. doi: 10.1212/01.wnl.0000194316.91908.8a. PMID 16434671
- [Background] Komatsu M, Waguri S, Chiba T, Murata S, Iwata J, Tanida I, Ueno T, Koike M, Uchiyama Y, Kominami E, Tanaka K. Loss of autophagy in the central nervous system causes neurodegeneration in mice. Nature. 2006 Jun 15;441(7095):880-4. doi: 10.1038/nature04723. Epub 2006 Apr 19. PMID 16625205
- [Background] Lattante S, de Calbiac H, Le Ber I, Brice A, Ciura S, Kabashi E. Sqstm1 knock-down causes a locomotor phenotype ameliorated by rapamycin in a zebrafish model of ALS/FTLD. Hum Mol Genet. 2015 Mar 15;24(6):1682-90. doi: 10.1093/hmg/ddu580. Epub 2014 Nov 19. PMID 25410659
- [Background] Lipton JO, Sahin M. The neurology of mTOR. Neuron. 2014 Oct 22;84(2):275-91. doi: 10.1016/j.neuron.2014.09.034. Epub 2014 Oct 22. PMID 25374355
- [Background] Mantovani S, Garbelli S, Pasini A, Alimonti D, Perotti C, Melazzini M, Bendotti C, Mora G. Immune system alterations in sporadic amyotrophic lateral sclerosis patients suggest an ongoing neuroinflammatory process. J Neuroimmunol. 2009 May 29;210(1-2):73-9. doi: 10.1016/j.jneuroim.2009.02.012. PMID 19307024
- [Background] Ravikumar B, Vacher C, Berger Z, Davies JE, Luo S, Oroz LG, Scaravilli F, Easton DF, Duden R, O'Kane CJ, Rubinsztein DC. Inhibition of mTOR induces autophagy and reduces toxicity of polyglutamine expansions in fly and mouse models of Huntington disease. Nat Genet. 2004 Jun;36(6):585-95. doi: 10.1038/ng1362. Epub 2004 May 16. PMID 15146184
- [Background] Shi CS, Shenderov K, Huang NN, Kabat J, Abu-Asab M, Fitzgerald KA, Sher A, Kehrl JH. Activation of autophagy by inflammatory signals limits IL-1beta production by targeting ubiquitinated inflammasomes for destruction. Nat Immunol. 2012 Jan 29;13(3):255-63. doi: 10.1038/ni.2215. PMID 22286270
- [Background] Staats KA, Hernandez S, Schonefeldt S, Bento-Abreu A, Dooley J, Van Damme P, Liston A, Robberecht W, Van Den Bosch L. Rapamycin increases survival in ALS mice lacking mature lymphocytes. Mol Neurodegener. 2013 Sep 11;8:31. doi: 10.1186/1750-1326-8-31. PMID 24025516
- [Background] Thomas M, Alegre-Abarrategui J, Wade-Martins R. RNA dysfunction and aggrephagy at the centre of an amyotrophic lateral sclerosis/frontotemporal dementia disease continuum. Brain. 2013 May;136(Pt 5):1345-60. doi: 10.1093/brain/awt030. Epub 2013 Mar 9. PMID 23474849
- [Background] Wang IF, Guo BS, Liu YC, Wu CC, Yang CH, Tsai KJ, Shen CK. Autophagy activators rescue and alleviate pathogenesis of a mouse model with proteinopathies of the TAR DNA-binding protein 43. Proc Natl Acad Sci U S A. 2012 Sep 11;109(37):15024-9. doi: 10.1073/pnas.1206362109. Epub 2012 Aug 29. PMID 22932872
- [Background] Zhang X, Li L, Chen S, Yang D, Wang Y, Zhang X, Wang Z, Le W. Rapamycin treatment augments motor neuron degeneration in SOD1(G93A) mouse model of amyotrophic lateral sclerosis. Autophagy. 2011 Apr;7(4):412-25. doi: 10.4161/auto.7.4.14541. Epub 2011 Apr 1. PMID 21193837
- [Derived] Trist BG, Fifita JA, Hogan A, Grima N, Smith B, Troakes C, Vance C, Shaw C, Al-Sarraj S, Blair IP, Double KL. Co-deposition of SOD1, TDP-43 and p62 proteinopathies in ALS: evidence for multifaceted pathways underlying neurodegeneration. Acta Neuropathol Commun. 2022 Aug 25;10(1):122. doi: 10.1186/s40478-022-01421-9. PMID 36008843